CLINICAL TRIAL: NCT04675359
Title: Comparison of the Treatment Results of Knee Osteoarthritis Using Adipose Tissue Mesenchymal Stromal Cells Derived Through Enzymatic Digestion and Mechanically Fragmented Adipose Tissue
Brief Title: Adipose-derived MSCs After Enzymatic Digestion vs. Mechanically Fragmented Fat Transfer in Knee Osteoarthritis Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSC
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Knee Osteoarthritis; Chondropathy
Keywords: MSC; SVF; adipose tissue; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Cartilage Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enzymatic digestion group (Active Comparator): A group treated with a stromal vascular fraction (SVF) with mesenchymal stromal cells (MSC) injection in the knee joint after an enzymatic digestion of autologous adipose tissue
  Interventions: Procedure: Autologous adipose derived Mesenchymal Stromal Cells (MSC) injection into the knee joint
- Mechanical fragmentation group (Active Comparator): A group treated with a mechanically fragmented (using Lipogems device) autologous adipose tissue injection in the knee joint
  Interventions: Procedure: Autologous adipose derived Mesenchymal Stromal Cells (MSC) injection into the knee joint

INTERVENTIONS:
Procedure: Autologous adipose derived Mesenchymal Stromal Cells (MSC) injection into the knee joint — Injections of the two adipose tissue derived products containing MSCs into the knee joints with osteoarthritis
  Other Names: Autologous mechanically fragmented adipose tissue injection into the knee joint using Lipogems device

SUMMARY:
The aim of the study is to compare the clinical effects of treatment of knee osteoarthritis using adipose tissue mesenchymal stromal cells obtained by an enzymatic method with the outcomes of the therapy with the mechanically fragmented adipose tissue. Identification and functional analysis of the regenerative capacity of MSCs derived from the adipose tissue depending on three variables (body weight, sex and age) will help to develop a targeted therapy for different groups of patients and will determine the effectiveness of both methods of treatment. An attempt was made to identify the groups of patients with the greatest regeneration potential of the adipose tissue, and thus indicate those with the most probable improvement of the joint condition.

DETAILED DESCRIPTION:
Based on the calculation of the sample size using power analysis of the test, investigators plan to include 100 adults with primary knee osteoarthritis in this study. The patients will undergo lipoaspiration under sterile conditions of the operating theatre, the collected lipoaspirates will be further processed - enzymatically with the use of collagenase or mechanically using the Lipogems system. After collection, lipoaspirates will be immediately transferred to the laboratory of the Department of Regenerative Medicine with a tissue and cells bank in Warsaw, and the preparations will be administered to the patients' knee joints in the operating room under ultrasound control.

The Lipogems system is defined as a minimal tissue manipulation system. In contrast, the administration of preparations produced using an enzymatic method requires advanced actions.

Lipoaspiration will be performed using blind cannulas and vacuum syringes introduced through the abdominal wall with a three-millimetre incision on the skin after previous injection to the adipose tissue with modified Klein's solution (500 ml of saline solution, 1 ml of adrenaline, 40 ml of 2% lignocaine), which makes the collection easier. 10 ml of the collected adipose tissue will be used to examine the samples after previous gradient drainage from Klein's solution. Immediately after collection, the samples will be sent to the laboratory for analysis (cell count testing, culture, phenotype identification, analysis by flow cytometry).

The patients will be monitored in the hospital outpatient clinic for one year after the procedure; the control visits will take place: after 2 and 6 weeks, then after 3 and 6 months and after a year. A physical examination and the assessment using the KOOS questionnaire will be performed. Before the procedure and after one year, an X-ray and MRI with T-2 Mapping will be carried out in order to evaluate the condition of the cartilage.

ELIGIBILITY:
Inclusion Criteria:

* Adults with symptomatic gonarthrosis diagnosed based on the X-ray, MRI and clinical examination, previously unsuccessfully treated (rehabilitation, NSAIDs, hyaluronic acid, platelet-rich plasma)
* Primary knee osteoarthritis
* Willingness and consent to participate in the study
* Readiness to attend control visits

Exclusion Criteria:

* Failure to meet the inclusion criteria
* Active chronic infection
* Metal implant made of a ferromagnetic material that will exclude the patient from magnetic resonance imaging
* Use of anticoagulants
* General and intra-articular use of steroids during the last year
* Pregnancy, breastfeeding
* Any autoimmune and rheumatic disease, or conditions that influence the accuracy of test results
* Taking drugs or cytostatic medications in the last 30 days
* Mental disorders, alcohol and drug addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in patients reported outcome measures - Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1,3,6 and 12 months after procedure
  The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life.The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included.
  Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Changes in flexibility of the knee joint | 1,3,6, and 12 months after procedure
  Range of motion assessment by goniometer measurements

SECONDARY OUTCOMES:
Changes in X-ray imaging of the knee joint in a standing position (AP view) | 6 months and 1 year after procedure
  Articular cartilage volume evaluation by joint gap measurements
Changes in MRI with T-2 Mapping of the knee cartilage | 6 months and 1 year after procedure
  Articular cartilage quality evaluation in T-2 Mapping

CONTACTS AND LOCATIONS:
Overall Officials: Artur Stolarczyk, MD, PhD, Principal Investigator — Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krzesniak AM, Radzimowski K, Stolarczyk A. Comparison of the treatment results of knee osteoarthritis using adipose tissue mesenchymal stromal cells derived through enzymatic digestion and mechanically fragmented adipose tissue. Medicine (Baltimore). 2021 Mar 5;100(9):e24777. doi: 10.1097/MD.0000000000024777. PMID 33655941